CLINICAL TRIAL: NCT07016438
Title: Phase I/IIa Clinical Study of PAL-222 Targeting Patients With Refractory Skin Ulcer
Brief Title: Clinical Study of PAL-222 Targeting Patients With Refractory Skin Ulcer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PharmaBio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAL-222-P3
Record Dates: First submitted 2025-05-08; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Refractory Skin Ulcer
MeSH Terms: conditions — Skin Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapeuitic group (Experimental)
  Interventions: Procedure: Transplant surgery

INTERVENTIONS:
Procedure: Transplant surgery — One piece of PAL-222 is implanted into the ulcer area through the surgical procedure.

SUMMARY:
The goal of this clinical trial is to assess safety and efficacy in patients with with Refractory skin ulcer no response to existing therapy.

The main measures it aims to answer are:

* Investigation of adverse events
* Changes in clinical testing data
* Changes in vital signs Participants will have one PAL-222 transplanted to the ulcer site. Researchers will compare before and after the transplantation to see if any safety issues are recognized.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients aged 20 years or older at the time of obtaining consent (2) Patients with skin ulcers whose ulcer size has decreased by less than 50% compared to before the start of treatment even after 4 weeks or more of conservative standard treatment (3) Patients with an ulcer of 1 cm2 or more and 3 cm2 or less after debridement (4) Patients with ulcers within 5 cm from the ulcer to be treated (5) Patients with no signs of local infection in the ulcer to be treated (6) If the ulcer had the bone exposure, it needs to be within 10% of the ulcer area (7) Patients with skin reflux pressure of 30 mmHg or more at the treatment site (if the patient has an ulcer on the lower leg or foot) (8) Patients who have received a written explanation of this clinical trial from the principal investigator or clinical investigator, fully understood the information, and given their own written consent to participate in this clinical trial (9) Patients who are able to follow oral or written instructions from the principal investigator or clinical investigator

Exclusion Criteria:

* (1) Patients with any of the following systemic diseases

  1. Poorly controlled diabetes mellitus (HbA1c greater than 10% at the most recent examination within 28 days prior to enrollment)
  2. Hypoalbuminemia (serum albumin level less than 2 g/dL)
  3. Patients requiring continuous oral steroids (prednisolone equivalent greater than 10 mg per day) (2) Patients requiring general anesthesia or lumbar anesthesia during the study period for the following reasons

  <!-- -->

  1. When local anesthesia is not appropriate for debridement due to scarring or hardness of the wound
  2. Patients who are mentally disturbed, have involuntary movements, or are unable to keep the wound at rest during transplantation (3) Patients with a history of allergy to human serum albumin, trypsin, anesthetics used in this study, antiseptics, or covering materials (4) Patients with abnormal findings on hematology, hematochemistry, coagulation, or urinalysis at the time of screening that would be problematic for participation in the clinical trial (5) Patients with positive HBs antigen, HCV antibody, HIV antibody, HTLV-1 antibody, or syphilis serology at screening (6) Patients with severe blood disorders (if any of the following criteria are met)

  <!-- -->

  1. Hemoglobin less than 10.0 g/dL
  2. White blood cell count less than 3,000 /microliter
  3. Neutrophil count less than 1,500 / microliter
  4. Platelet count less than 75,000 / microliter (7) Patients with severe heart failure (NYHA cardiac function classification III-IV) (8) Patients with severe hepatic impairment (with a history of or complicated by fulminant hepatitis, cirrhosis, liver tumor, or any of the following criteria)

  <!-- -->

  1. Total bilirubin 1.5x (upper limit of reference value) or higher
  2. AST (GOP) 3.0x (upper limit of reference value) or more
  3. ALT (GPT) 3.0x (upper limit of reference value) or more
  4. ALP 2.5x (upper limit of reference value) or higher (9) Patients with severe renal impairment (creatinine greater than 2 mg/dL) (10) Patients diagnosed with or requiring treatment for malignancy within 5 years prior to obtaining consent (11) Pregnant or lactating women, or patients who wish to become pregnant during the study period (12) Patients whose anticoagulant or antiplatelet medication cannot be discontinued prior to the clinical trial, as determined by the attending physician of the relevant department (13) Patients with drug addiction or alcoholism (14) Patients who are currently participating in another clinical trial (15) Patients who have participated in this clinical trial once and had PAL-222 implanted (16) Patients who are judged to be inappropriate as subjects by the investigator or subinvestigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The main measures it aims to answer safety. | 28days
  Safety Evaluation: Incidence, type, and severity of Adverse Events (AE)

CONTACTS AND LOCATIONS:
Locations (1):
- Kyoto University Hospital, Kyoto, Shogoin-kawahara-cho, Sakyo-ku, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: Undecided